CLINICAL TRIAL: NCT00929552
Title: Effect of n-3 LCPUFAs on Weight Reduction and Metabolic Syndrome.
Brief Title: Effect of Fish Oil on Markers of the Metabolic Syndrome in Overweight Adolescent Boys
Acronym: TeenFisk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D202; H-A-2007-0055
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome
Keywords: Blood pressure; Insulin sensitivity; Blood lipid profile
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Dietary Fats, Unsaturated; In Situ Hybridization, Fluorescence; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): Daily dose = 6g fish oil baked into rye bread and wheat rolls. Participants were asked to consume two slices of rye bread and one wheat roll pr day. The fish oil was micro-incapsulated.
  Interventions: Dietary Supplement: Dietary oils (fish, vegetable oil)
- Vegetable oil (Mix of canola, palm and soy oil) (Active Comparator): Daily dose = 6g vegetable oil baked into rye bread and wheat rolls. Participants were asked to consume two slices of rye bread and one wheat roll pr day.
  Interventions: Dietary Supplement: Dietary oils (fish, vegetable oil)

INTERVENTIONS:
Dietary Supplement: Dietary oils (fish, vegetable oil) — 6g pr day.

SUMMARY:
The aim of the study is to investigate if dietary fish oil has a beneficial effect on blood pressure, insulin sensitivity, blood lipid profile, body composition and metabolic rate in healthy, but slightly overweight, teenage boys.

We hypothesized that the n-3 long chain polyunsaturated fatty acids from fish oil might have greater effect during growth and development, as intervention trials studying the effect of fish oil on babies have shown greater effects than in adults.

ELIGIBILITY:
Inclusion Criteria:

* Weight above the 90th percentile for height and age.

Exclusion Criteria:

* Smoking, severe illnesses.

Ages: 13 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Markers of the metabolic syndrome. Blood pressure, insulin sensitivity, HDL-cholesterol and triacylglycerol. | Intervention period = 16 weeks

SECONDARY OUTCOMES:
Body composition | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Result] Pedersen MH, Molgaard C, Hellgren LI, Lauritzen L. Effects of fish oil supplementation on markers of the metabolic syndrome. J Pediatr. 2010 Sep;157(3):395-400, 400.e1. doi: 10.1016/j.jpeds.2010.04.001. Epub 2010 May 15. PMID 20472253